CLINICAL TRIAL: NCT01054131
Title: Peer to Peer Mentoring: Facilitating Individuals With Early Inflammatory Arthritis to Manage Their Arthritis: Peer Mentoring Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Arthritis Network (Network)
Responsible Party: Principal Investigator, Dr. Mary Bell, Rheumatologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Purpose: Supportive Care
Other Study IDs: 420-2009
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Early Inflammatory Arthritis; Chronic Disease
Keywords: peer support; peer mentor; self-management; early inflammatory arthritis; chronic disease
MeSH Terms: conditions — Arthritis; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: peer support — A quasi-experimental, before and after study design will obtain data for planning and implementing a larger-scale study. Exposures and outcomes will be measured at baseline, 3 months (immediate post 12-week program) and 6 months (3 months post-program). Ten individuals with EIA will be recruited by brief screening interviews to ensure they meet inclusion criteria. Each pair of peer mentor and EIA participant will meet at SHSC for an initial contact. EIA participants will receive informational, emotional and appraisal support from trained peer mentors by telephone or neutral private location at a time convenient for both parties, at least once a week for 12 weeks.

SUMMARY:
Inflammatory arthritis (IA) is a major cause of long-term disability. Peer support may be a solution to the common problem of delayed treatment. Early peer support may result in improved use of therapy, higher self-efficacy, reduced anxiety, and improved coping in the first two years post-diagnosis. The whole intervention study comprises of two parts: The first part involves the development and testing of a peer mentor training initiative, which is called "Peer to Peer Mentoring: Facilitating Individuals with Early Inflammatory Arthritis to Manage their Arthritis - Peer Mentor Training". The second part, which is the focus of this study, involves the delivery of a one-on-one peer support intervention from a trained peer mentor to an individual newly diagnosed with EIA. The feasibility and acceptability of the program will be determined, as well as the health outcomes following the participation of the program.

ELIGIBILITY:
Inclusion Criteria:

1. Have EIA disease duration within 6-52 weeks
2. At least 3 swollen joints, assessed by the treating rheumatologist, OR positive compression test for the metacarpophalangeal joints OR positive compression test for the metatarsophalangeal joints OR at least 30 minutes of morning stiffness
3. Prescription of a DMARD/biologic by the treating rheumatologist
4. Ability to speak and understand English without the aid of a secondary support person; AND
5. Capability to provide informed consent.

Exclusion Criteria:

1. IA disease duration less than 6 weeks or greater than 1 year
2. Previous or ongoing DMARD or biologic treatment
3. Inability to speak or read grade 6 English; AND
4. Inability to provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
DMARD adherence | 0, 3, 6 months

SECONDARY OUTCOMES:
coping efficacy | 0, 3 6 months
self-management | 0, 3, 6 months
anxiety | 0, 3, 6 months
self efficacy | 0, 3, 6 months
social support | 0, 3, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Bell, MD, FRCPC, Principal Investigator — Rheumatologist, Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Sandhu S, Veinot P, Embuldeniya G, Brooks S, Sale J, Huang S, Zhao A, Richards D, Bell MJ. Peer-to-peer mentoring for individuals with early inflammatory arthritis: feasibility pilot. BMJ Open. 2013 Mar 1;3(3):e002267. doi: 10.1136/bmjopen-2012-002267. PMID 23457326